CLINICAL TRIAL: NCT02738359
Title: Efficacy of Colonoscopy, Colon Capsule and Fecal Immunological Test for Colorectal Cancer Screening, in First Degree Relatives of Patients With Colorectal Neoplasia: a Prospective Randomized Study.
Brief Title: Efficacy of Colonoscopy, Colon Capsule and Fecal Immunological Test for Colorectal Cancer Screening
Acronym: FAMCAP
Status: Recruiting | Type: Observational
Sponsor: Hôpital Edouard Herriot (Other)
Collaborators: National Cancer Institute, France (Other Government); Medtronic (Industry)
Responsible Party: Principal Investigator, Jean Christophe Saurin, Professor, Hôpital Edouard Herriot
Other Study IDs: FAMCAP
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Colon Cancer; Rectum Cancer
Keywords: colon cancer; rectum cancer; colonoscopy; fecal immunological test; colon capsule
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1rst arm: optical colonoscopy (OC): t0: optical colonoscopy; Follow-up: yearly by phone call for three years
  Interventions: Procedure: optical colonoscopy
- 2nd arm: colon capsule endoscopy (CC): t0: colon capsule endoscopy -> if positive: OC; At three years: OC for those patients with negative initial CC; Follow-up: yearly by phone call for 3 years
  Interventions: Procedure: optical colonoscopy; Procedure: colon capsule endoscopy
- 3rd arm: fecal immunological test (FIT): FIT yearly for two years:
  t0: FIT -> if positive : OC; t = 1 year: FIT -> if positive : OC; t = 2 years: FIT -> if positive : OC; At three years: OC for those patients with negative FIT during the study Follow-up: yearly by phone call for 3 years
  Interventions: Procedure: optical colonoscopy; Diagnostic Test: fecal immunological test (FIT)

INTERVENTIONS:
Procedure: optical colonoscopy — optical colonoscopy
Procedure: colon capsule endoscopy — colon capsule endoscopy
  Groups: 2nd arm: colon capsule endoscopy (CC)
Diagnostic Test: fecal immunological test (FIT) — fecal immunological test (FIT)
  Groups: 3rd arm: fecal immunological test (FIT)

SUMMARY:
Efficacy of colonoscopy, colon capsule and fecal immunological test for colorectal cancer screening, in first degree relatives of patients with colorectal neoplasia: a prospective randomized study.

DETAILED DESCRIPTION:
Fecal immunological test (FIT) is the reference screening method in average risk patient. FIT is proposed every 2 years to all asymptomatic subjects with average risk aged from 50 to 74 years in France. Optical colonoscopy (OC) is the gold standard examination for patients at increased risk of colorectal cancer, like those with a first degree relative with colorectal cancer (relative risk between 2 and 4 times that of the general population). Colonoscopy should be performed in this high risk group before 50 years or 5 to 10 years before the earliest case of colorectal cancer. Optical colonoscopy has important limitations: complications (perforation, bleeding), need to use general anesthesia (in France 95% of colonoscopy are performed under general anesthesia), and low acceptability for screening even in high risk persons (40% in the best cases). In this high risk population, there is a potentially important place for alternative methods. FIT could be one of them, with already a significant amount of data suggesting its interest. No data are available in high risk French patients. Colon capsule endoscopy (CC) is a more recent technique with sparse data in this high risk group, and no prospective comparison with optical colonoscopy in this indication. Capsule endoscopy has the advantage of high feasibility, very low risk, probably (but to be demonstrated) increased acceptability, and represents the closest examination as compared to colonoscopy. This justifies a prospective study comparing in a randomized methodology these 3 modalities for the identification of advanced neoplastic lesions of the colon in well characterized group of subjects at high risk of colorectal cancer. The investigators propose a prospective, randomized protocol of non-inferiority in order to compare the two new strategies to the reference strategy for the detection of advanced colorectal neoplasia (colon or rectal cancers, large adenoma > 1 cm or high grade dysplasia ; 1st arm: OC first; 2nd arm: CC first, OC at 3 years for those patients with negative initial CC; 3rd arm: annual FIT for 2 years (t0, t = 1 year, t = 2 years), colonoscopy at 3 years for those patients with negative FIT during the study). The new strategies will be considered non-inferior to the reference strategy if the study allows to conclude that the absolute reduction of the proportion of detected patients is not greater than 3% in comparison to the reference strategy.

ELIGIBILITY:
Inclusion criteria:

* History of colorectal cancers (any age) in first-degree relatives (parents, children, siblings including half-brothers and sisters)
* Age > or = 45 years
* No previous colorectal cancer screening
* Informed patient
* Patient having signed the consent form
* Patient affiliated to a social security system or recipient of such system

Exclusion criteria:

* Any previous colorectal cancer screening:

  * History of blood tests in the stool (hemoccult, fecal immunological test, ...)
  * History of colonic capsule screening
  * History of colonoscopy
* Any known advanced neoplasia or colorectal cancer
* Known genetic predisposition to colorectal cancer (very high risk group)
* Adults protected by law (under guardianship or trusteeship)
* Other metastatic cancers
* Life-threatening diseases

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at high risk of colorectal cancer (first-degree relatives of patient with colorectal cancer) will be included prospectively in one of the 3 comparative arms.
Sampling Method: Probability Sample
Enrollment: 3250 (Estimated)
Dates: Start 2017-11-03 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence of advanced colorectal neoplasia or cancer identified by each screening strategy (OC, CC and FIT) | 3 years
  The main objective of the study is to compare two alternative methods (CC anf FIT) to OC in term of non-inferiority for the detection of advanced colorectal neoplasia (adenoma > 1 cm, adenoma with high grade dysplasia) or cancer. The method of the unilateral confidence interval of the difference will be used to test the non-inferiority. The strategies will be considered to be equivalent if the 95% confidence interval of the difference or the detection of advanced neoplasia won't exceed ±3%.

SECONDARY OUTCOMES:
Rate of colorectal cancer identified by each screening strategy | 3 years
  The rate of colorectal cancer identified by each strategy (= number of cancer identified by the strategy/number of patients for the strategy) will be calculated at the different steps of the study (t = first exam, t = yearly follow-up and/or interval colonoscopy, t = 3 years upon control colonoscopy) and over the full duration of the study. The rate of initial colorectal cancer, interval colorectal cancer, colorectal cancer at t=3 years and colorectal cancer identified over the duration of the study, respectively, have the same unit, i.e. the number of cancer identified by the strategy/number of patients for the strategy.

OTHER OUTCOMES:
Complication rate | 3 years
  Percentage of patient having experienced a significant complication from any screening strategy
Comparison of the strategies cost | 3 years
  Cumulative costs of each strategy compared to the detection of advanced neoplasia/cost per advanced neoplasia detected and cost/life-years gained.
Quality assessment of colonoscopy and capsule endoscopy | 3 years
  Quality assessment of colonoscopy and capsule endoscopy by analysing the rate of completion of colonoscopy and capsule endoscopy, and the caecal intubation rate.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Saurin, Pr, Principal Investigator — Hôpital Edouard Herriot - Hospices civils de Lyon; Robert Benamouzig, Pr, Study Chair — Hôpital Avicenne - Assistance publique-Hôpitaux de Paris
Locations (19):
- France (19):
  - CH Colmar, Colmar, Alsace
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Pessac, Aquitaine
  - Hôpital Edouard Herriot - Hospices civils de Lyon, Lyon, Auvergne-Rhône-Alpes
  - CHU de Saint-Etienne - Hôpital nord, Saint-Priest-en-Jarez, Auvergne-Rhône-Alpes
  - CHU de Dijon, Dijon, Bourgogne-Franche-Comté
  - CHU de Brest - Hôpital de la Cavale Blanche, Brest, Brittany Region
  - CHU de Rennes - Hôpital Pontchaillou, Rennes, Brittany Region
  - CHU de Besançon - Hôpital Minjoz, Besançon, Franche-Comté
  - CHU de Limoges - Hôpital Dupuytren, Limoges, Limousin
  - CHU de Toulouse, Toulouse, Midi-Pyrénées
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen, Normandy
  - CHU de Nantes - Hôpital de l'Hôtel-Dieu, Nantes, Pays de la Loire Region
  - CH d'Avignon, Avignon, Provence-Alpes-Côte d'Azur Region
  - Hôpital de la Timone - AP-HM, Marseille, Provence-Alpes-Côte d'Azur Region
  - CHU de Nice - Hôpital Archet II, Nice, Provence-Alpes-Côte d'Azure
  - Hôpital Avicenne - AP-HP, Bobigny, Île-de-France Region
  - CHI de Créteil, Créteil, Île-de-France Region
  - Hôpital Saint-Antoine - Assistance publique-Hôpitaux de Paris, Paris, Île-de-France Region
  - Hôpital Cochin - AP-HP, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT02738359/Prot_000.pdf